CLINICAL TRIAL: NCT04506801
Title: The Effect of Probiotics on Functional Constipation in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katarina Fehir Šola (Other)
Responsible Party: Sponsor-Investigator, Katarina Fehir Šola, Director of pharmacy, University of Zagreb
Organization: University of Zagreb (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 380-130/134-19-4
Record Dates: First submitted 2020-07-29; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Functional Constipation
Keywords: constipation; elderly; probiotics
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: randomised double-blind study
Who Masked: Care Provider
Masking Description: A randomization list will be generated by the permutated block method (variable size 4-6) and will be kept in a sealed envelope by a person not included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): liquid oral formulation 9 drops once a day
  Interventions: Other: Placebo
- Probiotic (Experimental): The probiotic contained Lactobacillus acidophilus LA3; 1 · 1011 CFU / g, Bifidobacterium animalis subsp. Lactis BLC1; 1.5 · 1011 CFU / g and Lactobacillus casei BGP93 2 · 1011cfu / g in the form of a liquid oral formulation
  Interventions: Dietary Supplement: Probalans senior

INTERVENTIONS:
Dietary Supplement: Probalans senior — Participants were told to consume 9 drops of study probiotics/placebo once a day for next 12-week intervention.
  Arms: Probiotic
Other: Placebo — Participants were told to consume 9 drops of study placebo one a day for the next 12-week intervention
  Arms: Placebo

SUMMARY:
The main scope of the proposed research in the framework is to investigate the effect of probiotic bacteria Lactobacillus acidophilus LA3, Bifidobacterium animalis ssp. lactis BLC1 i Lactobacillus casei BGP93 on functional constipation and on the quality of life of the elderly in a nursing home. The experimental part will consists of double-blind, placebo-controlled clinical trial over 12 weeks.

DETAILED DESCRIPTION:
During the first four weeks, the subjects were monitored primarily concerning bowel discharges and general health. After that initial four weeks, they are re-evaluated compliance with inclusion and exclusion criteria. Participants were allocated to the double-blind section of the trial (12 weeks), using o computer-generated to a placebo group or in the probiotic group in the form of a liquid oral formulation once a day. On first day of intervention participants provide a blood sample. All investigators, participants and study personnel were blinded to the order of randomization. Participants were told to consume 9 drops of study probiotics once a day for next 12-week intervention. On last day of intervention, participants provide a blood sample. The last four weeks of the double-blind section (week 9-12) participants an evaluation period in which the respondents were evaluated for the outcomes of the study. After completing the double-blind study, the participants were followed for an additional four weeks. Inclusive / Excluded criteria are evaluated on two occasions, at the time of inclusion in the 4-week introductory section and its end.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or more
* signed informed consent for study participation
* functional constipation defined by Rome IV criteria
* ability to understand the procedure

Exclusion Criteria:

* suspicion of obstructive ileus or previous obstructive ileus
* suspected or confirmed diagnosis: irritable colon syndrome, ulcerative colitis, Crohn's disease, malignant digestive tract disease
* diarrhoea of any cause within the last month
* acute infectious disease within the last month excluding people who use antibiotics
* persons who have opioid analgesics in pharmacotherapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Change in stool frequency in patients who use probiotics | 12 weeks
  The proportion of subjects who meet the criterion of "normal bowel movement" according to the Roman IV criteria, at least 3 times a week to no more than 3 times a day. This proportion will be determined for each of the 4 evaluation weeks and will be analyzed as a time-averaged proportion. The proportion will be estimated on the basis of the subjects' diaries in which, by days, with indicated dates, the subjects will record each bowel emptying. Investigators would inform the evidence base with regards to the multi-strained probiotic efficacy in treating constipation among the elderly.

SECONDARY OUTCOMES:
Change in hs-CRP at the blood of a patient who uses probiotics determined by immunoturbidimetric method | 12 weeks
  The secondary outcome is to investigate the effect of selected probiotic strains on the concentration of the marker of inflammation, hs c-reactive protein (hs-CRP) in the serum of the subjects. hs-CRP will be determined by the immunoturbidimetric method. Investigators wanted to study the effect of this multi-strained probiotic on clinical and laboratory parameters. Blood was collected before the probiotic intervention and after 12 weeks.
Change in glucose parameters of a patient who use probiotics determined by standard laboratory methods | 12 weeks
  Values of laboratory indicators - glucose metabolism will be monitored. Investigators wanted to study the effect of this multi-strained probiotic on glucose parameters. Blood was collected like in Outcome2, before the intervention and after the intervention.
Change in blood parameters- triglycerides of a patient who use probiotics determined by standard laboratory methods. | 12 weeks
  Values of laboratory indicators of lipid metabolism - triglycerides will be monitored. Blood was collected before and after the intervention. Investigators wanted to study the effect of multi-strain probiotics on triglycerides.
Change in blood parameter- total cholesterol of a patient determined by standard laboratory methods | 12 weeks
  Investigator monitoring change of laboratory indicators of total cholesterol in beginning and at the end of the intervention with multi-strain probiotics.
Change in HDL cholesterol in blood parameters of a patient who use probiotics determined by standard laboratory methods | 12 weeks
  Values of laboratory indicators of HDL (high density lipoprotein) will be monitoring during the intervention. Blood samples were collected before and after the intervention.
Change in LDL cholesterol at the blood of patients who use probiotics determined by standard laboratory methods | 12 weeks
  Investigator monitoring change of laboratory indicators of LDL(low density lipoprotein), before study and at the end of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Katarina Fehir Šola, Bjelovar, Croatia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication